CLINICAL TRIAL: NCT07169409
Title: Right Tools, Right Time, Right Place: Telehealth for Opioid Use Disorder in Vulnerable Settings
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boulder Care (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4R44DA061386 (NIH); 1R44DA061386-01 (NIH)
Record Dates: First submitted 2025-08-28; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
Keywords: telehealth
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Receiving Intervention (Experimental)
  Interventions: Drug: Telemedicine Buprenorphine Treatment

INTERVENTIONS:
Drug: Telemedicine Buprenorphine Treatment — With this NIDA-funded grant, the study team will identify app-based treatment workflows that are demonstrably effective in low-resource settings: namely, telehealth services that are accessible without high-speed internet and deliberately helping patients transition into OUD care from relevant health and community system settings. An intentional focus on rural areas and Black and Hispanic demographics will help enhance health equity, and support solutions for payors.

SUMMARY:
Our primary objective is to evaluate the ability of Boulder Care's telehealth-platform to create the necessary paradigmatic shift in Opioid Use Disorder (OUD) treatment to reach vulnerable populations, with targets that support both equitable and culturally-specific OUD treatment as well as business profitability.

ELIGIBILITY:
Inclusion Criteria:

* History of Opioid Use Disorder (OUD)
* Starting OUD treatment with buprenorphine, or within 45 days of starting or restarting this medication
* Speak and understand English

Exclusion Criteria:

* History of allergic reaction to buprenorphine
* Plans to move out of a Boulder Care-affiliated state site in the next 12 months (precluding continuation of care)
* Untreated mental or medical health conditions that, in the opinion of the participant, would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability, Appropriateness, Feasibility | 48 weeks
  To measure the participant intervention experience, the study team will utilize qualitative interview data with study participants. These data will be organized into the implementation science categories: Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM).
  The study team will determine whether each participant found the intervention to be feasible, acceptable, and/or appropriate. These findings will then be aggregated to better understand how participants experience the implementation of a telemedicine Opioid Use Disorder treatment organization, and will inform a future scaled-up implementation.

SECONDARY OUTCOMES:
CDC's Health-Related Quality of Life - 4 (CDC HRQOL-4, also called the "Healthy Days Measures") | 48 weeks
  Items include: self-rated health, physically unhealthy days, mentally unhealthy days, and activity limitation days.
  Values:
  Self-rated health: 1 = Excellent, 2 = Very good, 3 = Good, 4 = Fair, 5 = Poor → Minimum = 1 (Excellent), Maximum = 5 (Poor)
  Unhealthy days (physical/mental): Range 0-30 days in past 30 days
  → Minimum = 0, Maximum = 30
  Direction: Higher scores = worse outcomes (more unhealthy days or poorer self-rated health).
Brief Addiction Monitor | 48 weeks
  Description: A 17-item multidimensional measure covering three domains:
  1. Risk factors (e.g., substance use, craving, triggers)
  2. Protective factors (e.g., social support, confidence in recovery)
  3. Recovery environment (e.g., housing, employment, stress)
  Values:
  * Most items use a 0-30 day timeframe with counts (e.g. "How many days in the past 30 have you used alcohol?" → 0-30).
  * Some items use Likert-type 0-4 response options (e.g. "Not at all" to "Extremely").
  Scoring and Direction:
  * Higher scores on "risk" items = worse outcomes (e.g., more days using substances, more craving, more risk exposure).
  * Higher scores on "protective" items = better outcomes (e.g., greater confidence, more supportive contacts).
Visual Analogue Opioid Craving Scale | 48 weeks
  Description: A single-item measure where participants rate their current intensity of craving for opioids by marking a point along a straight line (100 mm in length). The left anchor indicates "No craving at all" and the right anchor indicates "Most intense craving imaginable".
  Values:
  Minimum = 0 mm (no craving at all) Maximum = 100 mm (most intense craving imaginable)
  Direction: Higher scores = worse outcome (greater opioid craving)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Baron, MPH, Study Director — Boulder Care
Locations (1):
- Boulder Care, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) from this study. Only aggregate study results will be reported.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459